CLINICAL TRIAL: NCT04158232
Title: Assessment of Regenerative Potential of Mature Permanent Teeth With Necrotic Pulps Using Two Revascularization Protocols. (In Vivo Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Ali, assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 306
Record Dates: First submitted 2019-10-31; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood clotting protocol for pulp regeneration (Active Comparator): pulp regeneration for mature teeth using blood clotting protocol
  Interventions: Other: Method
- platelet rich fibrin for pulp regeneration (Experimental): pulp regeneration for mature teeth using platelet rich fibrin (PRF)
  Interventions: Other: Method

INTERVENTIONS:
Other: Method — treatment of mature teeth with apical periodontitis

SUMMARY:
Regenerative endodontic procedures have been used to successfully treat human mature permanent teeth with necrotic pulps and apical periodontitis. Many researchers have begun to apply regenerative endodontic procedures to mature teeth in adult patients. Several clinical case reports have shown complete resolution of signs and symptoms of pulp necrosis in mature teeth, even those with large periapical lesions, as well as signs of pulp canal obliteration. thevaim of this study is To assess the regenerative potential of mature permanent teeth with necrotic pulps with platelet-rich fibrin (PRF) and blood clot using radiographic and clinical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mature teeth.
* Patients with periapical periodontitis.
* Maxillary anterior teeth only will be involved.
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
* Patients who will agree to the consent and will commit to follow up period.

Exclusion Criteria:

* Patients with immature roots.
* Patients with any systemic disease that may affect normal healing.
* Patients with swelling.
* Pregnant females.
* Patients who could/would not participate in a 1 year follow up.
* Patients with fistula.
* Patients with old age.
* Teeth with periodontal involvement.
* Teeth with vertical root fractures.
* Unrestorable teeth.

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-02 (Estimated); Primary Completion 2020-09-02 (Estimated); Study Completion 2020-11-02 (Estimated)

PRIMARY OUTCOMES:
clinical success | 9 months
  pulp vitality testing using electric pulp tester which detect response of pulp to electric current
radiographic success | 9 months
  healing of apical periodontitis by detecting change in apical radiolucency and absences of apical bone resorption

REFERENCES:
- [Derived] Youssef A, Ali M, ElBolok A, Hassan R. Regenerative endodontic procedures for the treatment of necrotic mature teeth: A preliminary randomized clinical trial. Int Endod J. 2022 Apr;55(4):334-346. doi: 10.1111/iej.13681. Epub 2022 Jan 31. PMID 35030270